CLINICAL TRIAL: NCT04192032
Title: Assessing the Effect of Flavor on College-Aged JUUL ENDS Users' Experiences and Exposures
Brief Title: Assessing the Effect of Flavor on ENDS Users' Experiences and Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Wasim Maziak, phd, Principal Investigator, Florida International University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 107308
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: In this study, we will recruit 80 young (18-24) JUUL users. Each participant will undergo 3 JUUL smoking sessions: 1) one where they will be vaping their preferred flavor; 2) one where they will be vaping the standard classic tobacco flavor; 3) a third one in which they will be vaping their preferred flavor in a JUUL Ecigarette (JEC) device that has a health warning label (HWL) attached to it. In addition, 10 participants will be invited to come back for two additional sessions: one in which they will be vaping their preferred flavor pod with a 3% nicotine concentration, and one in which they will use their preferred flavor pod with 0% nicotine concentration. Measurement of JUUL satisfaction, dependence, harm perception, and exposure to nicotine and toxicants will be conducted in all 5 sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Preferred flavor (5% nicotine) (Experimental): Preferred flavor Juul pod (5% nicotine)
  Interventions: Other: Preferred Juul pod flavor (5% nicotine)
- Classic Tobacco Flavor (Active Comparator): Control flavor (5% Classic Tobacco flavor Juul pod)
  Interventions: Other: Classic Tobacco Juul pod flavor (5% nicotine)
- Preferred flavor with HWL (Experimental): Preferred flavored Juul pod (5% nicotine) with HWL
  Interventions: Other: Preferred flavor with HWL
- Preferred flavor (3% nicotine) (Experimental): Preferred flavored Juul pod (3% nicotine)
  Interventions: Other: Preferred flavor, 3% nicotine
- Preferred flavor (0% nicotine) (Experimental): Preferred flavored Juul pod (0% nicotine)
  Interventions: Other: Preferred flavor, 0% nicotine

INTERVENTIONS:
Other: Preferred Juul pod flavor (5% nicotine) — Preferred Juul pod flavor (5% nicotine)
  Arms: Preferred flavor (5% nicotine)
Other: Classic Tobacco Juul pod flavor (5% nicotine) — Classic Tobacco Juul pod flavor (5% nicotine)
  Arms: Classic Tobacco Flavor
Other: Preferred flavor with HWL — Preferred flavor (5% nicotine) with HWL
  Arms: Preferred flavor with HWL
Other: Preferred flavor, 3% nicotine — Preferred flavor, 3% nicotine
  Arms: Preferred flavor (3% nicotine)
Other: Preferred flavor, 0% nicotine — Preferred flavor, 0% nicotine
  Arms: Preferred flavor (0% nicotine)

SUMMARY:
Recently, Maziak established a clinical lab at FIU to test the potential of waterpipe tobacco flavor regulation by the FDA. Given the importance of flavors on adolescent ENDS uptake and use, this lab is equipped to study the impact of flavor manipulations among adolescent ENDS users. In this study will recruit 80 young (18-24) JUUL users, in a 2x2 cross over lab study where in one condition they will use their JUUL preferred flavor and the other JUUL standard tobacco flavor. Our aims are to; Aim 1: Compare satisfaction, withdrawal suppression, and harm perception between tobacco-flavored and preferred flavor JUUL. This analysis will reveal the extent to which preferred flavor contributes to smoking satisfaction, withdrawal and craving suppression, and harm perception, compared to the standard tobacco flavor.

Aim 2: Compare puff topography and plasma nicotine levels between tobacco-flavored and preferred flavor JUUL. This analysis will examine the extent to which preferred flavor contributes to puffing behavior and toxicant exposure compared to the standard tobacco flavor.

Aim 3: Compare exhaled breath condensate (EBC) between tobacco-flavored and preferred flavor JUUL. This analysis will be the first to examine exposure to toxic aldehydes (formaldehyde, acetaldehyde, acrolein, benzaldehyde, and propionaldehyde) produced when using preferred flavor compared to the standard tobacco flavor.

Utilizing powerful clinical lab methods, this study will provide a broad testing of the effect of flavor manipulation on college-aged JUUL users, and provide experimental evidence about the potential of flavor-limitation policies on young ENDS users in the US.

DETAILED DESCRIPTION:
The use of e-cigarettes, or electronic nicotine delivery systems (ENDS), among adolescents and young adults continues to be a major public health issue. Because of appealing design, flavor selection, and popularity on social media, JUUL ENDS have gained popularity among young people, many of whom are not aware that JUUL devices contain nicotine. Regulating ENDS flavor represents a promising approach to curb ENDS use among US youth. This project will provide a broad testing of the effect of flavor manipulation on college-aged JUUL users, and assist public health authorities by providing answers to specific questions pertinent to the potential of ENDS regulation through flavor. These include: - How would flavor manipulation influence puffing behavior and plasma nicotine levels among JUUL smokers; - how would smoking smoking preferred or tobacco flavor reflects on smoker's satisfaction, withdrawal suppression, and harm perception; - how would flavor manipulation affect toxicant exposure levels measured on exhaled breath condensate (EBC) on JUUL smokers. Answers to these questions will help public health authorities predict the impact of flavor regulation on ENDS experimentation and continued use.

Recently, Maziak established a clinical lab at FIU to test the potential of waterpipe tobacco flavor regulation by the FDA. Given the importance of flavors on adolescent ENDS uptake and use, this lab is equipped to study the impact of flavor manipulations among adolescent ENDS users. In this study, we will recruit 80 young (18-24) JUUL users. Each participant will undergo 3 JUUL smoking sessions: 1) one where they will be vaping their preferred flavor; 2) one where they will be vaping the standard classic tobacco flavor; 3) a third one in which they will be vaping their preferred flavor in a JUUL Ecigarette (JEC) device that has a health warning label (HWL) attached to it. In addition, 10 participants will be invited to come back for two additional sessions: one in which they will be vaping their preferred flavor pod with a 3% nicotine concentration, and one in which they will use their preferred flavor pod with 0% nicotine concentration. Measurement of JUUL satisfaction, dependence, harm perception, and exposure to nicotine and toxicants will be conducted in all 5 sessions.

In the past few months, there has been an increasing number of reports of severe respiratory illness related to e-cigarette use. Both the U.S. Food and Drug Administration and the U.S. Centers for Disease Control and Prevention are currently investigating this outbreak. According to the CDC, these cases of e-cigarette, or vaping, associated lung injury (EVALI) have been reported in most patients that report a history of using THC-containing products, particularly those obtained off the street or from other informal sources (e.g. friends, family members, illicit dealers) (https://www.cdc.gov/tobacco/basic_information/e-cigarettes/severe-lung-disease.html). Several steps have been taken to minimize this risk (i.e., excluding marijuana and non-commercial vaping products users; excluding individuals with current potential EVALI symptoms; revision of the consent & re-consenting of participants that still need to complete study sessions; and providing all participants with a CDC fact sheet about EVALI). For further details please refer to the "Methods" & "Minimizing Risks" sections.

This study involves minimal risks (explained in more details below in section 8) to participants. These risks are: 1) JUUL use 2) Dependence 3) Venipuncture 4) EVALI risk. The risk involved in participating in the JUUL smoking sessions of this study will not exceed the risk that would otherwise be encountered during similar recreational sessions of JUUL smoking.

Participants will benefit by being involved in a study that can increase their awareness about the health and addictive consequences of JUUL smoking and they will be given educational materials at the end of the study that explain the health impact of e-cigarettes, the current EVALI outbreak, and include resources that are available to help with quitting such as national, state and local cessation services (please see the fact sheets attached in the methods section). The findings of this study will benefit the society at large. Understanding the effect of flavor manipulation on JUUL/ENDS users will be instrumental for local and federal health agencies' potential to curb the spread of ENDS use, and protect public health in the US.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals (determined by physical examination).
* Age of 18-24 years.
* Is willing to provide informed consent.
* Is willing to attend the lab as required by the study protocol.
* Regular Juul smokers (at least weekly for the past 3 months).
* Have abstained from Juul use for 12 hours prior to each session.

Exclusion Criteria:

* Report smoking cigarettes regularly (> 5 cigarettes/month in the past year).
* Report regular use of any other tobacco/nicotine product (e.g., e-cig, pipes, cigars) in the past year.
* Women who are breast-feeding or test positive for pregnancy (by urinalysis at screening).
* Individuals with self-reported history of chronic disease or psychiatric conditions.
* Individuals with history of or active cardiovascular disease, low or high blood pressure, seizures, and regular use of prescription medications (other than vitamins or birth control).

  * Individuals that report THC (marijuana) smoking/vaping.
  * Individuals that report the use of non-commercial (i.e., street) e-cigarette liquid or products
  * Individuals that report current EVALI-related symptoms (i.e., cough, shortness of breath, chest pain, nausea, vomiting, abdominal pain, diarrhea, fever, chills, or weight loss)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine | During five participant visits. Blood will be taken 2 times in each JUUL use session: before and after an approximately 60-min ad lib use period
  Change in plasma nicotine level

SECONDARY OUTCOMES:
Puff topography | During participants' five study visits. Puffing behavior is continuously measured during each Juul use session (an approximately 60-min ad lib use period)
  Measurement of puffing behavior
Minnesota Nicotine Withdrawal Scale | During participants' five study visits. Questionnaire will be administered 2 times in each Juul use session: before and after an approximately 60-min ad lib use period.]
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0 - 100. These items are presented as Visual Analog Scale with item (measure) centered above a horizontal line anchored on the left with not at all and on the right with extremely.
Tiffany-Drobes Questionnaire of Smoking Urges | During participants' five study visits. Questionnaire will be administered 2 times in each Juul use session: before and after an approximately 60-min ad lib use period.]
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 10 items that are scored 0 - 7. Rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Carbon monoxide levels | During participants' five study visits. Carbon monoxide levels will be measured 2 times in each Juul use session: before and after an approximately 60-min ad lib use period
  Change in carbon monoxide levels (in parts per million)
Harm perception | During participants' five study visits. Questionnaire will be administered after each of the 2 Juul use sessions. Each session is approximately 60-min ad lib use period.]
  This scale will assess waterpipe harm perception and measure perceptions of waterpipe relative risk compared to cigarettes. The scale will be scored on a 7-point scale ranging from 1 (not at all harmful), to 7 (extremely harmful).
Duke Sensory Questionnaire | During participants' five study visits. Questionnaire will be administered after each of the 2 smoking sessions. Each session is approximately 60-min ad lib use period.]
  This scale will assess participants sensory experience of the inhaled product. The scale has nine items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
The Cigarette/ENDS Evaluation Scale (WES) | During participants' five study visits. Questionnaire will be administered after each of the 2 Juul use sessions. Each session is approximately 60-min ad lib use period.
  This scale assesses participants' perception of ENDS use. The scale has 11 items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).

OTHER OUTCOMES:
Heart rate | During participants' five study visits. Heat rate will be measured from baseline continuously throughout each approximately 60-min session.
  Change in heart rate, measured in beats per minute
Blood pressure | During participants' five study visits. Blood pressure will be measured from baseline continuously throughout each approximately 60-min session
  Change in blood pressure, measured in mm/hg

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Maziak, MD, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No